CLINICAL TRIAL: NCT05415605
Title: Ultrasound Evaluation of Alveolar Stress by Measurement of Ultrasound Pleural Strain in Healthy Subjects
Acronym: LUNGSTRAIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: LOCAL/2019/LM-01; 2019-A01407-50 (Other: ANSM)
Record Dates: First submitted 2022-06-09; First posted 2022-06-13 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2022-08

CONDITIONS: Ultrasound Strain Measurement
Keywords: lung strain; speckle tracking; lung stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- healthy Volunteers (Experimental): Healthy male or female volunteers between 18 and 50 years old
  Interventions: Device: Lung Strain

INTERVENTIONS:
Device: Lung Strain — The main objective of this study is to describe the physiological values of lung strain in healthy volunteers as well as its variations induced by non-invasive positive pressure ventilation and their correlation with tidal volume.

SUMMARY:
In the critical patient, lung ultrasound is routinely performed for acute respiratory distress, adult respiratory distress syndrome and for hemodynamic evaluation. Its diagnostic performance is superior to that of chest radiography in the context of pleuropulmonary parenchymal pathologies. The search for lung sliding is performed to diagnose a pneumothorax or to search for the correct placement of the endotracheal intubation tube. However, this analysis is qualitative and is sometimes difficult to interpret. At present, there is no global evaluation technique at the patient's bed allowing to analyze simultaneously the alveolar recruitment, the pulmonary over-distension and the quality of the lung sliding, whereas the pulmonary damage is most often heterogeneous. The justification of our research project is based on the need to develop and validate a means of global and regional quantification of the mechanical and aeration properties of the lung parenchyma by the analysis of the acoustic markers of the pleura (pleural strain) by the ultrasound technique of speckle tracking. The aim is to establish the normal values of the pleural strain in healthy volunteers, in spontaneous ventilation and then in non-invasive mechanical ventilation, in order to vary the lung volume.

ELIGIBILITY:
Inclusion Criteria:

-Healthy volunteer male or female between 18 and 50 years old

Exclusion Criteria:

* History of traumatic or spontaneous pneumothorax
* History of connective tissue disease
* Any history of chronic respiratory disease
* Presence of an ongoing clinical respiratory Ear-Nose-Throat (ENT) or pulmonary syndrome (rhinitis, sinusitis, bronchitis, lung disease)
* History of gastro-duodenal reflux or stomach surgery

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-07-24 (Actual); Primary Completion 2022-07-27 (Actual); Study Completion 2022-07-27 (Actual)

PRIMARY OUTCOMES:
Lung Strain values | during the procedure (30 minutes)
  Lung strain values (%) in spontaneous ventilation and then under non-invasive mechanical ventilation (NIV) by varying tidal volume and PEEP

SECONDARY OUTCOMES:
Ultrasound semiology and normal values | during the procedure (30 minutes)
  Description of the ultrasound semiology and the normal values of the different strain parameters (Global longitudinal strain and strain rate) during apnea
Variations of the strain under NIV in the different pulmonary zones tested | during the procedure (30 minutes)
  Description of the variations of the strain and strain rate (inspiratory and expiratory) according to the variations of the level of inspiratory support and positive expiratory pressure (PEEP) under NIV in the different pulmonary zones tested
Longitudinal and transversal values of lung strain in the different pulmonary zones tested | during the procedure (30 minutes)
  Description of the longitudinal and transversal values of the lung strain and lung strain rate in the different pulmonary zones tested
Variations of the strain under NIV in the right ventricle | during the procedure (30 min)
  Description of the variations of the strain and strain rate (inspiratory and expiratory) according to the variations of the level of inspiratory support and positive expiratory pressure (PEEP) under NIV of the right ventricle
Variations of the strain under NIV of the diaphragm | during the procedure (30 minutes)
  Description of the variations of the strain and strain rate (inspiratory and expiratory) of the diaphragm according to the variations of the level of inspiratory support and positive expiratory pressure (PEEP) under NIV. The evaluation of the diaphragmatic strain will be coupled and compared to the fraction of shortening of the diaphragm, which is currently the ultrasound reference method to measure the function of this muscle

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nîmes, Hôpital Universitaire Carémeau, Nîmes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Duclos G, Marecal L, Resseguier N, Postzich M, Taguet C, Hraiech S, Leone M, Muller L, Zieleskiewicz L. Pleural lung sliding quantification using a speckle tracking technology: A feasibility study on 30 healthy volunteers. Comput Methods Programs Biomed. 2024 Sep;254:108316. doi: 10.1016/j.cmpb.2024.108316. Epub 2024 Jul 2. PMID 38968827